CLINICAL TRIAL: NCT03109795
Title: Anxiety-mediated Impairments in Large Elastic Artery Function and the Autonomic Nervous System
Acronym: ATLAS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding ended
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Gary L. Pierce, PhD, Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 201701762
Record Dates: First submitted 2017-04-04; First posted 2017-04-12 (Actual); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-06

CONDITIONS: Anxiety; Hypertension
MeSH Terms: conditions — Anxiety Disorders; Hypertension | interventions — Clonidine; Hydrochlorothiazide

STUDY DESIGN:
Intervention Model Description: Randomized, parallel, double-blind
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Clonidine (Experimental): To test the magnitude by which short-term (4 weeks) sympathetic nerve activity blockade (clonidine) improves large elastic artery stiffness, vascular inflammation and baroreflex function in subjects with moderate-to-high levels of anxiety
  Interventions: Drug: Clonidine Pill
- Hydrochlorothiazide (Active Comparator): Hydrochlorothiazide is a blood pressure-lowering control condition to compare to the effects of clonidine
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Clonidine Pill — sympathetic nerve activity blockade
  Arms: Clonidine
Drug: Hydrochlorothiazide — Blood pressure-lowering control condition
  Arms: Hydrochlorothiazide

SUMMARY:
The goal of this study is to evaluate the effectiveness of a short-term (4 weeks) pharmacological blockade of sympathetic nerve activity (clonidine) on anxiety symptoms, vascular function, inflammation, muscle sympathetic nerve activity, and oxidant stress in individuals with moderate-to-high anxiety. Individuals who are interested in the study will be identified by an online screening survey and will be contacted by the research team; advertisements, flyers and mass emails will direct individuals to the online screening survey. Those deemed eligible to participate will be randomized to either the clonidine intervention or hydrochlorothiazide as a blood-pressure lowering control condition. If eligible participants are currently being treated with blood pressure-lowering medications, they will be asked to go off these medications for 2 weeks prior to and during the course of the study. During the 2 week washout of blood pressure-lowering medications, participants will have safety visits (2 additional visits) that include measurements of blood pressure at 4 days and 7 days after the beginning of the washout period before the intervention. Assessments of anxiety symptoms via various surveys, vascular function (via non-invasive, well-established techniques), inflammation, muscle sympathetic nerve activity, and oxidant stress will be performed at baseline and at the post intervention session. Similar baseline measurements will be performed in control subjects with low or no anxiety for comparison, but these individuals will not undergo the intervention.

Participants with moderate-to-high anxiety will have a total of 6 visits to the laboratory, which includes the screening and consent (visit 1). Visit 2 (baseline measurements) and visit 6 (post-intervention measurements) will be more extensive (~4.5 hours) compared to the other visits (~30 min). Participants completing the washout will have an additional 2 visits (~30 min each) before "visit 2." Control subjects with low or no anxiety will only participate in visit 1 (screening and consent ) and visit 2 (baseline measurements).

DETAILED DESCRIPTION:
Anxiety disorders are the most common mental health problems in the United States, occurring in about 18% of adults per year, and a lifetime prevalence of approximately 28% (25). Importantly, anxiety disorders are associated with increased risk for sudden cardiac death and non-fatal myocardial infarction (27, 46) independent of other mood disorders (13, 15). However, establishing a clear consensus on the mechanism(s) by which chronic anxiety confers cardiovascular disease (CVD) risk has proven difficult. Previous studies examining the potential role of vascular dysfunction in subjects with anxiety have been confounded by co-morbidities (e.g., hypertension, smoking, obesity) (31, 38) and added psychiatric disorders (63). Additionally, studies focusing on the relation between anxiety and robust predictors of CVD mortality, such as large elastic artery (e.g., aortic, carotid) stiffness, have been lacking.

Anxiety is experienced as negative feelings of threat, restlessness, tension and irritability, and somatic symptoms, such as palpitations, sweating, trembling, and dry mouth (57). Patients with clinically diagnosed anxiety disorder demonstrate more than 2-fold increase in future CVD events (23). Despite the strong association between anxiety and CVD risk, there is currently a gap in knowledge describing potential mechanisms by which anxiety leads to CVD. Evidence suggests that chronically high levels of anxiety may be associated with the progression of subclinical atherosclerosis such as carotid artery intima-media thickness (38) and elevated inflammation (5, 44). Symptoms of anxiety may also lead to impairment in resistance vessel dilator function (53). However, few studies have examined large elastic artery stiffness in subjects with high levels of anxiety. This is clinically important because large elastic artery stiffness (i.e., carotid and aortic) is a robust independent risk factor for CVD events such as stroke and myocardial infarction (6, 19, 59, 61). Interestingly, greater large elastic artery stiffness (aortic) is observed with higher resting muscle sympathetic nerve activity (MSNA) in healthy individuals even after adjusting for BP (9, 55). In this regard, numerous studies have shown that high MSNA independent of any increase in blood pressure can have deleterious vascular (7, 17, 32), metabolic (2, 20), cardiac (50, 52), and renal effects (1, 14, 54). Higher tonic MSNA is an independent determinant of aortic artery stiffness as assessed by the gold standard carotid-femoral pulse wave velocity (PWV) in healthy humans (55). Even acute increases in MSNA, such as during mental stress which is a potent stimulus for increases in MSNA (3), can lead to transiently greater large elastic artery stiffness (40). Furthermore, in healthy humans, acute mental stress induces transient endothelial dysfunction (16), an important modulator of arterial stiffness. Given findings from previous studies (22) showing that anxiety symptoms are associated with indices of elevated sympathetic nerve activity (e.g., elevated circulating norepinephrine), lead us to our overall hypothesis that anxiety-induced sympathetic overactivity leads to increased large elastic artery (carotid and aortic) stiffness in subjects with chronic anxiety.

The purpose of this study is to 1) determine the extent to which measures of vascular and autonomic function (large elastic artery stiffness, vascular inflammation and baroreflex function) is impaired in subjects with moderate-to-high anxiety, and 2) test the magnitude by which short-term (4 weeks) sympathetic nerve activity blockade (clonidine) improves large elastic artery stiffness, vascular inflammation and baroreflex function in subjects with moderate-to-high levels of anxiety.

In healthy subjects, chronic anxiety has been associated with increased risk of cardiac events (13, 15, 23). Interestingly, evidence suggests baroreflex function is reduced in subjects with anxiety (48, 60), thus adding additional cardiac risk burden to this population. Consistent with this, impairment in cardiac baroreflex sensivity (BRS) is a significant predictor of cardiac arrhythmias and myocardial infarction mortality (29, 56). Moreover, reduced cardiac BRS is a sensitive predictor of mortality after myocardial infarction (28, 30), particularly in subjects with anxiety (47). Reduced baroreflex activation can be attributed, in part, to reduced distensibility of baroreceptor regions within the elastic carotid and aortic arteries as a result of increased arterial stiffness (8). Given the associated risk of cardiac BRS impairment with anxiety, and the increase in large elastic artery stiffness in this population, there is a critical need to examine whether reductions in SNA and large elastic artery stiffness ameliorates cardiac BRS impairment in subjects with anxiety, thus providing experimental support for the novel idea that anxiety leads to increased CVD risk at least in part through elevated large artery stiffness.

ELIGIBILITY:
Inclusion Criteria for participants with moderate-to-high anxiety to undergo drug intervention:

* Willing and able to provide written, signed consent after the nature of the study has been explained, and prior to any research-related procedures.

Age is > or = 18 and < or = 79 years

No history of cardiovascular disease (e.g., heart attack, stroke, heart failure, valvular heart disease, cardiomyopathy), or peripheral arterial disease.

Non-smokers, defined as no history of smoking or no smoking for at least the past 3 months.

Normal resting 12-lead ECG (no evidence of myocardial infarction, left ventricular hypertrophy, left-bundle branch block, 2nd or 3rd degree AV block, atrial fibrillation/flutter, atherosclerosis).

Blood chemistries indicative of normal renal (creatinine <2.0mg/dl), liver (<3 times upper limit for ALT, AST), and thyroid function (TSH between 0.4 - 5.0 mU/L) or on stable thyroid medication with no dose change for 3 months.

Exclusion Criteria:

* Current use of clonidine or beta-blockers

Current use of antihypertensive medications for reasons other than hypertension (e.g., hydrochlorothiazide for leg edema or kidney stone prevention, beta-blockers for tremor)

Difficult to control hypertension (e.g., on 2 or 3 antihypertensive medications)

Low blood pressure (e.g., systolic BP < 110 mmHg)

Hypertensive and have not been stable on their current antihypertensive medication regimen for at least 6 months

Blood pressure not controlled either on or off antihypertensive medications (e.g., BP > 150/100)

Current diagnosis or history of cancer, liver disease, HIV/AIDS

History of brain tumor, aneurysm or injury

Clinical diagnosis of mental health disorders such as bipolar disorder or schizophrenia

History of cardiovascular disease such as heart angioplasty/stent or bypass surgery, myocardial infarction, stroke, heart failure with or without LV ejection fraction <40%, cardiomyopathy, valvular heart disease, cardiomyopathy, heart transplantation, atherosclerosis.

Current tobacco user or history of tobacco use within the past 3 months (cigarettes, cigars, chewing tobacco, Hookah).

History of lung emphysema, chronic bronchitis or chronic obstructive pulmonary disease (COPD).

Abnormal resting 12-lead ECG (e.g., evidence of myocardial infarction, left ventricular hypertrophy, left-bundle branch block, 2nd or 3rd degree AV block, atrial fibrillation/flutter, atherosclerosis).

Serious neurologic disorders including seizures.

History of renal failure, dialysis or kidney transplant.

Use of any investigational products or investigational medical devices within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.

Recent flu-like symptoms within the past 2 weeks.

Pregnant or breastfeeding at screening, or planning to become pregnant (self or partner) at any time during the study. A urinary pregnancy test will be done on all females. If test is positive, the subject will be excluded.

History of rheumatoid arthritis, Grave's disease, systemic lupus erythamatosis, and Wegener's granulomatosis.

Taking anticoagulation, anti-seizure, or antipsychotic agents.

Start of or dose change to an antidepressant or anti-anxiety medication within the past 3 months (if no change in medication or dose in past 3 month, then subject will be eligible).

Immunodeficiency or systemic autoimmune disease.

History of bleeding disorders or conditions of the microcirculation (i.e. von Willebrand disease, Raynaud's disease).

History of co-morbid condition that would limit life expectancy to <1 year.

Taking chronic non-steroidal anti-inflammatory drugs (NSAIDs) such as aspirin, indomethacin, naproxen, acetaminophen (Tylenol®), ibuprofen (Advil®, Motrin®) and not able or willing to go off of for 2 weeks prior to each study visit.

Taking cox-2 inhibitors (Celebrex®, Vioxx®, etc) or allopurinol (Zyloprim®, Lopurin®, Aloprim®).

Taking steroids or biologics: corticosteroids (prednisone); methotrexate, infliximib (Remicade®), etaneracept (Enbrel®); anakinra (Kineret®).

Those who are currently donating blood, platelets, or plasma at the time of screening.

Vulnerable populations (prisoners, etc.) will not be eligible to participate in this study.

On weight loss drugs (i.e. orilistat (Xenical®), sibutramine (Meridia®), phenylpropanol-amine (Acutrim®)), or similar over-the-counter medications within 3 months of screening.

Any surgery within 30 days of screening

Those who currently donate blood, platelets, or plasma

Any condition that, in the view of the PI or Co-I, places the subject at high risk or poor treatment and study compliance.

We will also enroll 36 participants ages 18-79 years (50% men, 50% women) with low or no anxiety as control subjects to participate in only baseline testing (not participate in the drug intervention).

Inclusion criteria:

Willing and able to provide written, signed consent after the nature of the study has been explained, and prior to any research-related procedures.

Age is > or = 18 and < or = 79 years

No history of cardiovascular disease (e.g., heart attack, stroke, heart failure, valvular heart disease, cardiomyopathy), or peripheral arterial disease.

Non-smokers, defined as no history of smoking or no smoking for at least the past 3 months.

Normal resting 12-lead ECG (no evidence of myocardial infarction, left ventricular hypertrophy, left-bundle branch block, 2nd or 3rd degree AV block, atrial fibrillation/flutter, atherosclerosis).

Blood chemistries indicative of normal renal (creatinine <2.0mg/dl), liver (<3 times upper limit for ALT, AST), and thyroid function (TSH between 0.4 - 5.0 mU/L) or on stable thyroid medication with no dose change for 3 months.

Exclusion Criteria:

Current use of clonidine or beta-blockers

Current use of antihypertensive medications for reasons other than hypertension (e.g., hydrochlorothiazide for leg edema or kidney stone prevention, beta-blockers for tremor)

Difficult to control hypertension (e.g., on 2 or 3 antihypertensive medications)

Low blood pressure (e.g., systolic BP < 110 mmHg)

Hypertensive and have not been stable on their current antihypertensive medication regimen for at least 6 months

Blood pressure not controlled either on or off antihypertensive medications (e.g., BP > 150/100)

Current diagnosis or history of cancer, liver disease, HIV/AIDS

History of brain tumor, aneurysm or injury

Clinical diagnosis of mental health disorders such as bipolar disorder or schizophrenia

History of cardiovascular disease such as heart angioplasty/stent or bypass surgery, myocardial infarction, stroke, heart failure with or without LV ejection fraction <40%, cardiomyopathy, valvular heart disease, cardiomyopathy, heart transplantation, atherosclerosis.

Current tobacco user or history of tobacco use within the past 3 months (cigarettes, cigars, chewing tobacco, Hookah).

History of lung emphysema, chronic bronchitis or chronic obstructive pulmonary disease (COPD).

Abnormal resting 12-lead ECG (e.g., evidence of myocardial infarction, left ventricular hypertrophy, left-bundle branch block, 2nd or 3rd degree AV block, atrial fibrillation/flutter, atherosclerosis).

Serious neurologic disorders including seizures.

History of renal failure, dialysis or kidney transplant.

Use of any investigational products or investigational medical devices within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.

Recent flu-like symptoms within the past 2 weeks.

Pregnant or breastfeeding at screening, or planning to become pregnant (self or partner) at any time during the study. A urinary pregnancy test will be done on all females. If test is positive, the subject will be excluded.

History of rheumatoid arthritis, Grave's disease, systemic lupus erythamatosis, and Wegener's granulomatosis.

Taking anticoagulation, anti-seizure, or antipsychotic agents.

Start of or dose change to an antidepressant or anti-anxiety medication within the past 3 months (if no change in medication or dose in past 3 month, then subject will be eligible).

Immunodeficiency or systemic autoimmune disease.

History of bleeding disorders or conditions of the microcirculation (i.e. von Willebrand disease, Raynaud's disease).

History of co-morbid condition that would limit life expectancy to <1 year.

Taking chronic non-steroidal anti-inflammatory drugs (NSAIDs) such as aspirin, indomethacin, naproxen, acetaminophen (Tylenol®), ibuprofen (Advil®, Motrin®) and not able or willing to go off of for 2 weeks prior to each study visit.

Taking cox-2 inhibitors (Celebrex®, Vioxx®, etc) or allopurinol (Zyloprim®, Lopurin®, Aloprim®).

Taking steroids or biologics: corticosteroids (prednisone); methotrexate, infliximib (Remicade®), etaneracept (Enbrel®); anakinra (Kineret®).

Those who are currently donating blood, platelets, or plasma at the time of screening.

Vulnerable populations (prisoners, etc.) will not be eligible to participate in this study.

On weight loss drugs (i.e. orilistat (Xenical®), sibutramine (Meridia®), phenylpropanol-amine (Acutrim®)), or similar over-the-counter medications within 3 months of screening.

Any surgery within 30 days of screening

Those who currently donate blood, platelets, or plasma

Any condition that, in the view of the PI or Co-I, places the subject at high risk or poor treatment and study compliance.

We will also enroll 36 participants ages 18-79 years (50% men, 50% women) with low or no anxiety as control subjects to participate in only baseline testing (not participate in the drug intervention). These subjects will be either lean (body mass index < 25) or on the obesity spectrum (body mass index > 30).

Because obesity is linked with hypertension and type 2 diabetes, enrollment of subjects may include those with pre-hypertension or hypertension (systolic blood pressure >/= 120 - <180 mmHg- average of at least 3 measurements 2 min apart after 10 min seated resting position), and/or pre-diabetes (defined as fasting blood glucose between 100-126 mg/dl, fasting blood glucose of 140-199 mg/dl at 120 min of an oral glucose tolerance test, or HbA1C of 6-6.5%) or type 2 diabetes (defined as fasting blood glucose between >126 mg/dl, fasting blood glucose of >199 mg/dl at 120 min of an oral glucose tolerance test, or HbA1C > 6.5%). These subjects may be taking anti-hypertensive and/or diabetes (anti-hyperglycemic) medications. Subjects will be asked to refrain from medications the morning of the study visit, and to bring their medications with them to take immediately following their study visit.

Inclusion criteria:

Willing and able to provide written, signed consent after the nature of the study has been explained, and prior to any research-related procedures.

Age is > or = 18 and < or = 79 years

No history of cardiovascular disease (e.g., heart attack, stroke, heart failure, valvular heart disease, cardiomyopathy), or peripheral arterial disease.

Non-smokers, defined as no history of smoking or no smoking for at least the past 3 months.

Normal resting 12-lead ECG (no evidence of myocardial infarction, left ventricular hypertrophy, left-bundle branch block, 2nd or 3rd degree AV block, atrial fibrillation/flutter, atherosclerosis).

Blood chemistries indicative of normal renal (creatinine <2.0mg/dl), liver (<3 times upper limit for ALT, AST), and thyroid function (TSH between 0.4 - 5.0 mU/L) or on stable thyroid medication with no dose change for 3 months.

Exclusion Criteria:

Current diagnosis or history of cancer, liver disease, HIV/AIDS

History of brain tumor, aneurysm or injury

Clinical diagnosis of mental health disorders such as bipolar disorder or schizophrenia

History of cardiovascular disease such as heart angioplasty/stent or bypass surgery, myocardial infarction, stroke, heart failure with or without LV ejection fraction <40%, cardiomyopathy, valvular heart disease, cardiomyopathy, heart transplantation, atherosclerosis.

Current tobacco user or history of tobacco use within the past 3 months (cigarettes, cigars, chewing tobacco, Hookah).

History of lung emphysema, chronic bronchitis or chronic obstructive pulmonary disease (COPD).

Abnormal resting 12-lead ECG (e.g., evidence of myocardial infarction, left ventricular hypertrophy, left-bundle branch block, 2nd or 3rd degree AV block, atrial fibrillation/flutter, atherosclerosis).

Serious neurologic disorders including seizures.

History of renal failure, dialysis or kidney transplant.

Use of any investigational products or investigational medical devices within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.

Recent flu-like symptoms within the past 2 weeks.

Pregnant or breastfeeding at screening, or planning to become pregnant (self or partner) at any time during the study. A urinary pregnancy test will be done on all females. If test is positive, the subject will be excluded.

History of rheumatoid arthritis, Grave's disease, systemic lupus erythamatosis, and Wegener's granulomatosis.

Taking anticoagulation, anti-seizure, or antipsychotic agents.

Start of or dose change to an antidepressant or anti-anxiety medication within the past 3 months (if no change in medication or dose in past 3 month, then subject will be eligible).

Immunodeficiency or systemic autoimmune disease.

History of bleeding disorders or conditions of the microcirculation (i.e. von Willebrand disease, Raynaud's disease).

History of co-morbid condition that would limit life expectancy to <1 year.

Taking chronic non-steroidal anti-inflammatory drugs (NSAIDs) such as aspirin, indomethacin, naproxen, acetaminophen (Tylenol®), ibuprofen (Advil®, Motrin®) and not able or willing to go off of for 2 weeks prior to each study visit.

Taking cox-2 inhibitors (Celebrex®, Vioxx®, etc) or allopurinol (Zyloprim®, Lopurin®, Aloprim®).

Taking steroids or biologics: corticosteroids (prednisone); methotrexate, infliximib (Remicade®), etaneracept (Enbrel®); anakinra (Kineret®).

Those who are currently donating blood, platelets, or plasma at the time of screening.

Vulnerable populations (prisoners, etc.) will not be eligible to participate in this study.

On weight loss drugs (i.e. orilistat (Xenical®), sibutramine (Meridia®), phenylpropanol-amine (Acutrim®)), or similar over-the-counter medications within 3 months of screening.

Any surgery within 30 days of screening

Those who currently donate blood, platelets, or plasma

Any condition that, in the view of the PI or Co-I, places the subject at high risk or poor treatment and study compliance.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth W Holwerda, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amann K, Rump LC, Simonaviciene A, Oberhauser V, Wessels S, Orth SR, Gross ML, Koch A, Bielenberg GW, VAN Kats JP, Ehmke H, Mall G, Ritz E. Effects of low dose sympathetic inhibition on glomerulosclerosis and albuminuria in subtotally nephrectomized rats. J Am Soc Nephrol. 2000 Aug;11(8):1469-1478. doi: 10.1681/ASN.V1181469. PMID 10906160
- [Background] Anderson EA, Hoffman RP, Balon TW, Sinkey CA, Mark AL. Hyperinsulinemia produces both sympathetic neural activation and vasodilation in normal humans. J Clin Invest. 1991 Jun;87(6):2246-52. doi: 10.1172/JCI115260. PMID 2040704
- [Background] Anderson EA, Wallin BG, Mark AL. Dissociation of sympathetic nerve activity in arm and leg muscle during mental stress. Hypertension. 1987 Jun;9(6 Pt 2):III114-9. doi: 10.1161/01.hyp.9.6_pt_2.iii114. PMID 3596778
- [Background] Arch JJ, Wolitzky-Taylor KB, Eifert GH, Craske MG. Longitudinal treatment mediation of traditional cognitive behavioral therapy and acceptance and commitment therapy for anxiety disorders. Behav Res Ther. 2012 Aug;50(7-8):469-78. doi: 10.1016/j.brat.2012.04.007. Epub 2012 May 7. PMID 22659156
- [Background] Bankier B, Barajas J, Martinez-Rumayor A, Januzzi JL. Association between C-reactive protein and generalized anxiety disorder in stable coronary heart disease patients. Eur Heart J. 2008 Sep;29(18):2212-7. doi: 10.1093/eurheartj/ehn326. Epub 2008 Jul 4. PMID 18603621
- [Background] Ben-Shlomo Y, Spears M, Boustred C, May M, Anderson SG, Benjamin EJ, Boutouyrie P, Cameron J, Chen CH, Cruickshank JK, Hwang SJ, Lakatta EG, Laurent S, Maldonado J, Mitchell GF, Najjar SS, Newman AB, Ohishi M, Pannier B, Pereira T, Vasan RS, Shokawa T, Sutton-Tyrell K, Verbeke F, Wang KL, Webb DJ, Willum Hansen T, Zoungas S, McEniery CM, Cockcroft JR, Wilkinson IB. Aortic pulse wave velocity improves cardiovascular event prediction: an individual participant meta-analysis of prospective observational data from 17,635 subjects. J Am Coll Cardiol. 2014 Feb 25;63(7):636-646. doi: 10.1016/j.jacc.2013.09.063. Epub 2013 Nov 13. PMID 24239664
- [Background] Bevan RD. Trophic effects of peripheral adrenergic nerves on vascular structure. Hypertension. 1984 Nov-Dec;6(6 Pt 2):III19-26. doi: 10.1161/01.hyp.6.6_pt_2.iii19. PMID 6394491
- [Background] Bruno RM, Ghiadoni L, Seravalle G, Dell'oro R, Taddei S, Grassi G. Sympathetic regulation of vascular function in health and disease. Front Physiol. 2012 Jul 24;3:284. doi: 10.3389/fphys.2012.00284. eCollection 2012. PMID 22934037
- [Background] Casey DP, Curry TB, Joyner MJ, Charkoudian N, Hart EC. Relationship between muscle sympathetic nerve activity and aortic wave reflection characteristics in young men and women. Hypertension. 2011 Mar;57(3):421-7. doi: 10.1161/HYPERTENSIONAHA.110.164517. Epub 2011 Jan 17. PMID 21242459
- [Background] Chapleau MW, Cunningham JT, Sullivan MJ, Wachtel RE, Abboud FM. Structural versus functional modulation of the arterial baroreflex. Hypertension. 1995 Aug;26(2):341-7. doi: 10.1161/01.hyp.26.2.341. PMID 7543454
- [Background] Dindo L, Recober A, Marchman JN, Turvey C, O'Hara MW. One-day behavioral treatment for patients with comorbid depression and migraine: a pilot study. Behav Res Ther. 2012 Sep;50(9):537-43. doi: 10.1016/j.brat.2012.05.007. Epub 2012 May 27. PMID 22728646
- [Background] Fairfax ST, Padilla J, Vianna LC, Davis MJ, Fadel PJ. Spontaneous bursts of muscle sympathetic nerve activity decrease leg vascular conductance in resting humans. Am J Physiol Heart Circ Physiol. 2013 Mar 1;304(5):H759-66. doi: 10.1152/ajpheart.00842.2012. Epub 2013 Jan 4. PMID 23292718
- [Background] Fiedorowicz JG, He J, Merikangas KR. The association between mood and anxiety disorders with vascular diseases and risk factors in a nationally representative sample. J Psychosom Res. 2011 Feb;70(2):145-54. doi: 10.1016/j.jpsychores.2010.07.010. Epub 2010 Sep 18. PMID 21262417
- [Background] Fisher JP, Young CN, Fadel PJ. Central sympathetic overactivity: maladies and mechanisms. Auton Neurosci. 2009 Jun 15;148(1-2):5-15. doi: 10.1016/j.autneu.2009.02.003. Epub 2009 Mar 6. PMID 19268634
- [Background] Frasure-Smith N, Lesperance F. Depression and anxiety as predictors of 2-year cardiac events in patients with stable coronary artery disease. Arch Gen Psychiatry. 2008 Jan;65(1):62-71. doi: 10.1001/archgenpsychiatry.2007.4. PMID 18180430
- [Background] Ghiadoni L, Donald AE, Cropley M, Mullen MJ, Oakley G, Taylor M, O'Connor G, Betteridge J, Klein N, Steptoe A, Deanfield JE. Mental stress induces transient endothelial dysfunction in humans. Circulation. 2000 Nov 14;102(20):2473-8. doi: 10.1161/01.cir.102.20.2473. PMID 11076819
- [Background] Grassi G, Giannattasio C, Failla M, Pesenti A, Peretti G, Marinoni E, Fraschini N, Vailati S, Mancia G. Sympathetic modulation of radial artery compliance in congestive heart failure. Hypertension. 1995 Aug;26(2):348-54. doi: 10.1161/01.hyp.26.2.348. PMID 7635545
- [Background] Grassi G, Turri C, Seravalle G, Bertinieri G, Pierini A, Mancia G. Effects of chronic clonidine administration on sympathetic nerve traffic and baroreflex function in heart failure. Hypertension. 2001 Aug;38(2):286-91. doi: 10.1161/01.hyp.38.2.286. PMID 11509491
- [Background] Hansen TW, Staessen JA, Torp-Pedersen C, Rasmussen S, Li Y, Dolan E, Thijs L, Wang JG, O'Brien E, Ibsen H, Jeppesen J. Ambulatory arterial stiffness index predicts stroke in a general population. J Hypertens. 2006 Nov;24(11):2247-53. doi: 10.1097/01.hjh.0000249703.57478.78. PMID 17053547
- [Background] Hausberg M, Mark AL, Hoffman RP, Sinkey CA, Anderson EA. Dissociation of sympathoexcitatory and vasodilator actions of modestly elevated plasma insulin levels. J Hypertens. 1995 Sep;13(9):1015-21. doi: 10.1097/00004872-199509000-00012. PMID 8586819
- [Background] Holwerda SW, Reynolds LJ, Restaino RM, Credeur DP, Leidy HJ, Thyfault JP, Fadel PJ. The influence of reduced insulin sensitivity via short-term reductions in physical activity on cardiac baroreflex sensitivity during acute hyperglycemia. J Appl Physiol (1985). 2015 Dec 15;119(12):1383-92. doi: 10.1152/japplphysiol.00584.2015. Epub 2015 Oct 15. PMID 26472870
- [Background] Hughes JW, Watkins L, Blumenthal JA, Kuhn C, Sherwood A. Depression and anxiety symptoms are related to increased 24-hour urinary norepinephrine excretion among healthy middle-aged women. J Psychosom Res. 2004 Oct;57(4):353-8. doi: 10.1016/j.jpsychores.2004.02.016. PMID 15518669
- [Background] Janszky I, Ahnve S, Lundberg I, Hemmingsson T. Early-onset depression, anxiety, and risk of subsequent coronary heart disease: 37-year follow-up of 49,321 young Swedish men. J Am Coll Cardiol. 2010 Jun 29;56(1):31-7. doi: 10.1016/j.jacc.2010.03.033. PMID 20620714
- [Background] A-Tjak JG, Davis ML, Morina N, Powers MB, Smits JA, Emmelkamp PM. A meta-analysis of the efficacy of acceptance and commitment therapy for clinically relevant mental and physical health problems. Psychother Psychosom. 2015;84(1):30-6. doi: 10.1159/000365764. Epub 2014 Dec 24. PMID 25547522
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Knight RG, Waal-Manning HJ, Spears GF. Some norms and reliability data for the State--Trait Anxiety Inventory and the Zung Self-Rating Depression scale. Br J Clin Psychol. 1983 Nov;22 (Pt 4):245-9. doi: 10.1111/j.2044-8260.1983.tb00610.x. PMID 6640176
- [Background] Kubzansky LD, Cole SR, Kawachi I, Vokonas P, Sparrow D. Shared and unique contributions of anger, anxiety, and depression to coronary heart disease: a prospective study in the normative aging study. Ann Behav Med. 2006 Feb;31(1):21-9. doi: 10.1207/s15324796abm3101_5. PMID 16472035
- [Background] La Rovere MT, Bigger JT Jr, Marcus FI, Mortara A, Schwartz PJ. Baroreflex sensitivity and heart-rate variability in prediction of total cardiac mortality after myocardial infarction. ATRAMI (Autonomic Tone and Reflexes After Myocardial Infarction) Investigators. Lancet. 1998 Feb 14;351(9101):478-84. doi: 10.1016/s0140-6736(97)11144-8. PMID 9482439
- [Background] La Rovere MT, Pinna GD, Maestri R, Sleight P. Clinical value of baroreflex sensitivity. Neth Heart J. 2013 Feb;21(2):61-3. doi: 10.1007/s12471-012-0349-8. PMID 23184601
- [Background] La Rovere MT, Specchia G, Mortara A, Schwartz PJ. Baroreflex sensitivity, clinical correlates, and cardiovascular mortality among patients with a first myocardial infarction. A prospective study. Circulation. 1988 Oct;78(4):816-24. doi: 10.1161/01.cir.78.4.816. PMID 3168190
- [Background] Lambert E, Dawood T, Straznicky N, Sari C, Schlaich M, Esler M, Lambert G. Association between the sympathetic firing pattern and anxiety level in patients with the metabolic syndrome and elevated blood pressure. J Hypertens. 2010 Mar;28(3):543-50. doi: 10.1097/HJH.0b013e3283350ea4. PMID 20139772
- [Background] Mancia G, Giannattasio C, Grassi G. Arterial distensibility in cardiovascular diseases. J Nephrol. 1998 Nov-Dec;11(6):284-8. PMID 10048493
- [Background] Muzi M, Goff DR, Kampine JP, Roerig DL, Ebert TJ. Clonidine reduces sympathetic activity but maintains baroreflex responses in normotensive humans. Anesthesiology. 1992 Nov;77(5):864-71. doi: 10.1097/00000542-199211000-00005. PMID 1443738
- [Background] Newsom SA, Richards JC, Johnson TK, Kuzma JN, Lonac MC, Paxton RJ, Rynn GM, Voyles WF, Bell C. Short-term sympathoadrenal inhibition augments the thermogenic response to beta-adrenergic receptor stimulation. J Endocrinol. 2010 Sep;206(3):307-15. doi: 10.1677/JOE-10-0152. Epub 2010 Jul 5. PMID 20603265
- [Background] Padilla J, Young CN, Simmons GH, Deo SH, Newcomer SC, Sullivan JP, Laughlin MH, Fadel PJ. Increased muscle sympathetic nerve activity acutely alters conduit artery shear rate patterns. Am J Physiol Heart Circ Physiol. 2010 Apr;298(4):H1128-35. doi: 10.1152/ajpheart.01133.2009. Epub 2010 Feb 12. PMID 20154260
- [Background] Parati G, Di Rienzo M, Bertinieri G, Pomidossi G, Casadei R, Groppelli A, Pedotti A, Zanchetti A, Mancia G. Evaluation of the baroreceptor-heart rate reflex by 24-hour intra-arterial blood pressure monitoring in humans. Hypertension. 1988 Aug;12(2):214-22. doi: 10.1161/01.hyp.12.2.214. PMID 3410530
- [Background] Parati G, Saul JP, Di Rienzo M, Mancia G. Spectral analysis of blood pressure and heart rate variability in evaluating cardiovascular regulation. A critical appraisal. Hypertension. 1995 Jun;25(6):1276-86. doi: 10.1161/01.hyp.25.6.1276. PMID 7768574
- [Background] Paterniti S, Zureik M, Ducimetiere P, Touboul PJ, Feve JM, Alperovitch A. Sustained anxiety and 4-year progression of carotid atherosclerosis. Arterioscler Thromb Vasc Biol. 2001 Jan;21(1):136-41. doi: 10.1161/01.atv.21.1.136. PMID 11145945
- [Background] Peltonen GL, Scalzo RL, Schweder MM, Larson DG, Luckasen GJ, Irwin D, Hamilton KL, Schroeder T, Bell C. Sympathetic inhibition attenuates hypoxia induced insulin resistance in healthy adult humans. J Physiol. 2012 Jun 1;590(11):2801-9. doi: 10.1113/jphysiol.2011.227090. Epub 2012 Apr 10. PMID 22495590
- [Background] Phillips AA, Bredin SS, Cote AT, Drury CT, Warburton DE. Aortic distensibility is reduced during intense lower body negative pressure and is related to low frequency power of systolic blood pressure. Eur J Appl Physiol. 2013 Mar;113(3):785-92. doi: 10.1007/s00421-012-2489-3. Epub 2012 Sep 14. PMID 22971725
- [Background] Pierce GL, Casey DP, Fiedorowicz JG, Seals DR, Curry TB, Barnes JN, Wilson DR, Stauss HM. Aortic pulse wave velocity and reflecting distance estimation from peripheral waveforms in humans: detection of age- and exercise training-related differences. Am J Physiol Heart Circ Physiol. 2013 Jul 1;305(1):H135-42. doi: 10.1152/ajpheart.00916.2012. Epub 2013 Apr 26. PMID 23624628
- [Background] Pierce GL, Donato AJ, LaRocca TJ, Eskurza I, Silver AE, Seals DR. Habitually exercising older men do not demonstrate age-associated vascular endothelial oxidative stress. Aging Cell. 2011 Dec;10(6):1032-7. doi: 10.1111/j.1474-9726.2011.00748.x. Epub 2011 Oct 17. PMID 21943306
- [Background] Pierce GL, Lesniewski LA, Lawson BR, Beske SD, Seals DR. Nuclear factor-kappaB activation contributes to vascular endothelial dysfunction via oxidative stress in overweight/obese middle-aged and older humans. Circulation. 2009 Mar 10;119(9):1284-92. doi: 10.1161/CIRCULATIONAHA.108.804294. Epub 2009 Feb 23. PMID 19237660
- [Background] Pitsavos C, Panagiotakos DB, Papageorgiou C, Tsetsekou E, Soldatos C, Stefanadis C. Anxiety in relation to inflammation and coagulation markers, among healthy adults: the ATTICA study. Atherosclerosis. 2006 Apr;185(2):320-6. doi: 10.1016/j.atherosclerosis.2005.06.001. Epub 2005 Jul 11. PMID 16005881
- [Background] Powers MB, Zum Vorde Sive Vording MB, Emmelkamp PM. Acceptance and commitment therapy: a meta-analytic review. Psychother Psychosom. 2009;78(2):73-80. doi: 10.1159/000190790. Epub 2009 Jan 14. PMID 19142046
- [Background] Roest AM, Martens EJ, de Jonge P, Denollet J. Anxiety and risk of incident coronary heart disease: a meta-analysis. J Am Coll Cardiol. 2010 Jun 29;56(1):38-46. doi: 10.1016/j.jacc.2010.03.034. PMID 20620715
- [Background] Roest AM, Martens EJ, Denollet J, de Jonge P. Prognostic association of anxiety post myocardial infarction with mortality and new cardiac events: a meta-analysis. Psychosom Med. 2010 Jul;72(6):563-9. doi: 10.1097/PSY.0b013e3181dbff97. Epub 2010 Apr 21. PMID 20410247
- [Background] Sanchez-Gonzalez MA, Guzik P, May RW, Koutnik AP, Hughes R, Muniz S, Kabbaj M, Fincham FD. Trait anxiety mimics age-related cardiovascular autonomic modulation in young adults. J Hum Hypertens. 2015 Apr;29(4):274-80. doi: 10.1038/jhh.2014.72. Epub 2014 Aug 28. PMID 25355009
- [Background] Saul JP, Rea RF, Eckberg DL, Berger RD, Cohen RJ. Heart rate and muscle sympathetic nerve variability during reflex changes of autonomic activity. Am J Physiol. 1990 Mar;258(3 Pt 2):H713-21. doi: 10.1152/ajpheart.1990.258.3.H713. PMID 2316686
- [Background] Sen S, Young D. Effect of sodium deprivation on cardiac hypertrophy in spontaneously hypertensive rats: influence of aging. J Mol Cell Cardiol. 1991 Jun;23(6):695-704. doi: 10.1016/0022-2828(91)90979-v. PMID 1834855
- [Background] Silver AE, Christou DD, Donato AJ, Beske SD, Moreau KL, Magerko KA, Seals DR. Protein expression in vascular endothelial cells obtained from human peripheral arteries and veins. J Vasc Res. 2010;47(1):1-8. doi: 10.1159/000231715. Epub 2009 Aug 6. PMID 19672102
- [Background] Simpson P. Norepinephrine-stimulated hypertrophy of cultured rat myocardial cells is an alpha 1 adrenergic response. J Clin Invest. 1983 Aug;72(2):732-8. doi: 10.1172/JCI111023. PMID 6135712
- [Background] Stillman AN, Moser DJ, Fiedorowicz J, Robinson HM, Haynes WG. Association of anxiety with resistance vessel dysfunction in human atherosclerosis. Psychosom Med. 2013 Jul-Aug;75(6):537-44. doi: 10.1097/PSY.0b013e31829a0ae3. Epub 2013 Jun 20. PMID 23788697
- [Background] Strojek K, Grzeszczak W, Gorska J, Leschinger MI, Ritz E. Lowering of microalbuminuria in diabetic patients by a sympathicoplegic agent: novel approach to prevent progression of diabetic nephropathy? J Am Soc Nephrol. 2001 Mar;12(3):602-605. doi: 10.1681/ASN.V123602. PMID 11181810
- [Background] Swierblewska E, Hering D, Kara T, Kunicka K, Kruszewski P, Bieniaszewski L, Boutouyrie P, Somers VK, Narkiewicz K. An independent relationship between muscle sympathetic nerve activity and pulse wave velocity in normal humans. J Hypertens. 2010 May;28(5):979-84. doi: 10.1097/hjh.0b013e328336ed9a. PMID 20408258
- [Background] Thayer JF, Lane RD. The role of vagal function in the risk for cardiovascular disease and mortality. Biol Psychol. 2007 Feb;74(2):224-42. doi: 10.1016/j.biopsycho.2005.11.013. Epub 2006 Dec 19. PMID 17182165
- [Background] Tyrer P, Baldwin D. Generalised anxiety disorder. Lancet. 2006 Dec 16;368(9553):2156-66. doi: 10.1016/S0140-6736(06)69865-6. PMID 17174708
- [Background] Vallbo AB, Hagbarth KE, Torebjork HE, Wallin BG. Somatosensory, proprioceptive, and sympathetic activity in human peripheral nerves. Physiol Rev. 1979 Oct;59(4):919-57. doi: 10.1152/physrev.1979.59.4.919. No abstract available. PMID 227005
- [Background] van Sloten TT, Sedaghat S, Laurent S, London GM, Pannier B, Ikram MA, Kavousi M, Mattace-Raso F, Franco OH, Boutouyrie P, Stehouwer CDA. Carotid stiffness is associated with incident stroke: a systematic review and individual participant data meta-analysis. J Am Coll Cardiol. 2015 Nov 10;66(19):2116-2125. doi: 10.1016/j.jacc.2015.08.888. PMID 26541923
- [Background] Victor RG, Leimbach WN Jr. Effects of lower body negative pressure on sympathetic discharge to leg muscles in humans. J Appl Physiol (1985). 1987 Dec;63(6):2558-62. doi: 10.1152/jappl.1987.63.6.2558. PMID 3436888
- [Background] Virtanen R, Jula A, Salminen JK, Voipio-Pulkki LM, Helenius H, Kuusela T, Airaksinen J. Anxiety and hostility are associated with reduced baroreflex sensitivity and increased beat-to-beat blood pressure variability. Psychosom Med. 2003 Sep-Oct;65(5):751-6. doi: 10.1097/01.psy.0000088760.65046.cf. PMID 14508016
- [Background] Vlachopoulos C, Aznaouridis K, Stefanadis C. Prediction of cardiovascular events and all-cause mortality with arterial stiffness: a systematic review and meta-analysis. J Am Coll Cardiol. 2010 Mar 30;55(13):1318-27. doi: 10.1016/j.jacc.2009.10.061. PMID 20338492
- [Background] Westen D, Morrison K. A multidimensional meta-analysis of treatments for depression, panic, and generalized anxiety disorder: an empirical examination of the status of empirically supported therapies. J Consult Clin Psychol. 2001 Dec;69(6):875-99. PMID 11777114
- [Background] Yeragani VK, Tancer M, Seema KP, Josyula K, Desai N. Increased pulse-wave velocity in patients with anxiety: implications for autonomic dysfunction. J Psychosom Res. 2006 Jul;61(1):25-31. doi: 10.1016/j.jpsychores.2005.10.011. PMID 16813842

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clonidine | Hydrochlorothiazide
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated before any participants were randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Clonidine | Hydrochlorothiazide | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Aortic Stiffness
Description: Aortic stiffness as determined by the carotid-femoral pulse wave velocity technique
Time Frame: 4 weeks
Population: Study was terminated before any participant was randomized to groups.
Arm/Group | Clonidine | Hydrochlorothiazide
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Study terminated before randomization
Description: Study terminated before randomization
Arm/Group | Clonidine | Hydrochlorothiazide
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study was terminated before any participants were randomized because of lack of funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT03109795/Prot_SAP_000.pdf